CLINICAL TRIAL: NCT05633797
Title: The Occurrence of Atrial Fibrillation After Totally Endoscopic Cardiac Surgery
Acronym: AFMICS-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After the passing of the principal investigator, the clinical trial could not be continued.
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: f/2022/127
Record Dates: First submitted 2022-11-18; First posted 2022-12-01 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: Postoperative atrial fibrillation; Minimally invasive cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Totally endoscopic cardiac surgery (Experimental): Patients will be monitored using the FibriCheck application to detect atrial fibrillation until 30 days postoperative.
  Interventions: Device: FibriCheck

INTERVENTIONS:
Device: FibriCheck — During the patient's intensive care unit (ICU) stay, they will be monitored constantly to detect atrial fibrillation (standard care). After ICU dismissal, patients will be monitored using the FibriCheck application to detect atrial fibrillation until 30 days postoperative. Patients need to use the FibriCheck application for a minimum of 3x/day and can perform extra measurements when symptoms are present.

SUMMARY:
The aim of this study is to investigate the occurrence of new-onset postoperative atrial fibrillation after totally endoscopic cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Patients undergoing elective endoscopic cardiac surgery (totally endoscopic coronary artery bypass grafting or endoscopic valve replacement)

Exclusion Criteria:

* Preoperative atrial fibrillation
* Patients that do not understand Dutch or French or English
* Patients that do not have a smartphone
* Concomitant or redo surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
The occurence of new-onset postoperative atrial fibrillation using constant electrocardiogram monitoring and photoplethysmography (FibriCheck) | Until 30 days postoperatively
  New-onset postoperative atrial fibrillation will be detected until 30 days postoperatively. Constant electrocardiogram monitoring is performed at the intensive care unit (ICU). After dismissal from the ICU, the FibriCheck application is used to detect atrial fibrillation using photoplethysmography. Patients need to use the application three times a day and when symptoms are present.

SECONDARY OUTCOMES:
The effect of the closure of the pericardium on the development of new-onset postoperative atrial fibrillation | Intraoperative
  It will be registered if the pericardium is closed unilateral, bilateral or left open.

CONTACTS AND LOCATIONS:
Overall Officials: Alaaddin Yilmaz, MD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No